CLINICAL TRIAL: NCT05908942
Title: Comparison of the Efficacy of Genicular Nerve Phenol Ablation and Radiofrequency Ablation for Pain Management in Patients With Knee Osteoarthritis
Brief Title: Genicular RFT vs Phenol Management in Patients With Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, medical doctor, Diskapi Teaching and Research Hospital
Other Study IDs: Genicular
Record Dates: First submitted 2023-06-05; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Knee Pain Chronic
Keywords: Genicular radiofrequency; Phenol; Pain treatment; Osteoarthritis
MeSH Terms: conditions — Agnosia; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- RF group: 32 patients with knee osteoarthritis to undergo radiofrequency treatment of genicular nerves
  Interventions: Device: Nerve ablation
- Phenol group: 32 patients with knee osteoarthritis to undergo phenol treatment of genicular nerves
  Interventions: Device: Nerve ablation

INTERVENTIONS:
Device: Nerve ablation — radiofrequency and phenol ablation of the genicular nerves will be performed

SUMMARY:
The aim of this study was to compare the efficacy of phenol and radiofrequency ablation for genicular nerve neurolysis in severe knee pain. The invesigators compare the efficacy of radiofrequency and phenol applications on numerical pain score and Western Ontario and McMaster Universi- ties Osteoarthritis Index (WOMAC) before, 1 and 3 months after the procedure. The procedures will be performed by applying radiofrequency waves and phenol to the genicular nerves under ultrasound guidance.

DETAILED DESCRIPTION:
Ultrasound-guided genicular nerve ablation is a minimally invasive procedure that reduces or eliminates pain in patients with knee pain by destroying the nerves that transmit pain with heat or chemical drugs such as phenol. Genicular nerve ablation is an effective treatment option for patients with chronic knee pain who cannot undergo prosthesis surgery. In this method, radiofrequency waves or phenol are applied to the nerves going to the knee joint, preventing the transmission of pain signals to the brain.

The procedure is applied as follows:

Haemodynamic monitoring is provided. Superomedial genicular nerve (SMGS), superolateral genicular nerve (SLGS), inferomedial genicular nerve (IMGS) are the nerves to be blocked. The 8-12 Hz linear ultrasound probe is first placed superomedial to the knee and the SMGS and genicular artery are visualised at the junction of the shaft and condyle of the femur. The skin is locally anaesthetised with 2% lidocaine (2 cc) and the needle is inserted in plane with the ultrasound probe. For radiofrequency ablation The cannula placed close to the nerve is connected to the radiofrequency generator with the help of cables. At the tip of the needle, 2% lidocaine (1 cc) is administered and the nerve is heated by applying radiofrequency current. Ablation is performed at 80 °C for 1 minute. This procedure is repeated for other genicular nerves. For phenol ablation, 1 mL of 7% phenol solution is applied to cause neurolysis with the help of a needle placed close to the nerve. Phenol provides ablation by denaturing the proteins in the structure of the nerve.

Patients will be evaluated on NRS and WOMAC scales before, 1 and 3 months after the procedure. The evaluation will be done face to face and by telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe knee pain due to knee osteoarthritis (0-10 pain of intensity 6 and above on an inter-numeric pain scale)
* Permanent pain for more than 6 months
* Grade 3 or 4 in the radiological Kellgren-Lawrence classification having osteoarthritis
* Pain with conservative methods such as analgesics and physiotherapy treatment failure

Exclusion Criteria:

* History of intra-articular knee intervention in the last 6 months
* Cognitive impairment
* Hepatic or renal insufficiency
* Severe psychiatric illness
* Local or systemic infection
* Coagulopathy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Genicular nerve radiofrequency and phenol for knee osteoarthritis
  male and female patients undergoing ablation
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Change from Baseline NRS at 3 months
  Patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity.
Western Ontario and McMaster Universi- ties Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 3 months
  The WOMAC Pain score ranges from 0 to 20 with higher scores equating to greater pain with activities of daily living. The generic pain scale ranges from 0 to 10 for the OAI and 0 to 100 for MOST, with higher scores equating to greater pain

CONTACTS AND LOCATIONS:
Overall Officials: Gevher R Genç Perdecioğlu, Study Chair — Diskapi TRH
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara, Yenimahalle
  - Diskapi Training and Research Hospital, Ankara